CLINICAL TRIAL: NCT00044564
Title: An Uncontrolled Phase II, Multi Center Trial Evaluating Antitumor Efficacy and Safety of Bay 59-8862 in Patients With Advanced Renal Cell Carcinoma
Brief Title: Evaluation of Bay 59-8862 in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100386
Record Dates: First submitted 2002-08-30; First posted 2002-09-04 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: Taxane; Renal Cell Carcinoma; Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — IDN 5109

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Bay 59-8862

INTERVENTIONS:
Drug: Bay 59-8862 — 75 mg/m2 of BAY 59-8862 intravenously over one hour. Treatment will be repeated once every 3 weeks and tumor measurements will be made every 2 cycles till progression, unacceptable toxicity or consent withdrawal

SUMMARY:
In patients with renal cell cancer, most frequent methods of treatment include surgery, chemotherapy, hormonal therapy, and immunotherapy. Renal cell carcinoma is usually considered to be radioresistant and chemoresistant. In patients with metastatic disease, the options are limited. The taxanes are among the most commonly used class of chemotherapy agents in clinical oncology today but they are not effective in renal cancers; the development of Bay 59-8862 targets taxane-resistant tumors and the current protocol is designed to test the safety and efficacy of Bay 59-8862 in patients with advanced renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria: - measurable disease as defined by the presence of at least one measurable lesion - prior immunotherapy (up to 2 regimens) or prior radiotherapy is permitted but at least 4 weeks must have elapsed prior to enter study - life expectancy of at least 12 weeks - adequate bone marrow, liver and kidney function Exclusion Criteria: - excluded medical conditions like: pre-existing neuropathy, active heart diseases or ischemia, serious infections, HIV infection, chronic hepatitis B or C, brain metastasis, seizures, hypersensitivity to taxanes, organ transplants, some previous cancers - excluded therapies and medications, previous and concomitant such as: anticancer chemotherapy or immunotherapy during the study or within 4 weeks prior to study entry; more than two prior anticancer chemotherapy regimens; radiotherapy during study or within 4 weeks prior to study entry; bone marrow transplant - others: pregnant or breast-feeding patients; both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial; substance abuse, medical, psychological or social conditions that may interfere with the patient's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2001-12; Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Objective overall tumor response rate calculated as the percentage of patients with complete and partial responses | At baseline and every 2 cycles during the treatment period

SECONDARY OUTCOMES:
Duration of response | At baseline and every cycle during the treatment period
Overall survival | Till end of follow up period (up to 2 years)
Time to progression | Throughout study
Pharmacokinetics assessment | At cycle 1
Qualitative and quantitative toxicity profile | Day 1 of each cycle or as clinically indicated
Physical examinations | As clinically indicated
Vital signs data | Throughout study period
Abnormal laboratory tests | Prior to every cycle till last study visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (27):
- United States (12):
  - La Jolla, California
  - Muncie, Indiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Greenbelt, Maryland
  - Detroit, Michigan
  - Southfield, Michigan
  - St Louis, Missouri
  - Billings, Montana
  - New Brunswick, New Jersey
  - Salt Lake City, Utah
  - Milwaukee, Wisconsin
- Canada (3):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Greater Sudbury, Ontario
- France (2):
  - Caen
  - Montpellier
- Germany (5):
  - Heidelberg, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Düsseldorf, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
- Rotterdam, Netherlands
- United Kingdom (4):
  - Plymouth, Devon
  - Manchester, Greater Manchester
  - Cardiff, South Glamorgan
  - Sutton, Surrey